CLINICAL TRIAL: NCT02330978
Title: Intravitreal Autologous Bone Marrow-derived Mesenchymal Stem Cell Transplantation in Patients With Advanced Glaucoma. Phase I: Safety Study.
Brief Title: Intravitreal Mesenchymal Stem Cell Transplantation in Advanced Glaucoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, JAYTER SILVA DE PAULA, Associate Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRP 14151/2010
Record Dates: First submitted 2014-12-31; First posted 2015-01-05 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Retinal Degeneration; Primary Open-angle Glaucoma
MeSH Terms: conditions — Retinal Degeneration; Glaucoma, Open-Angle | interventions — Culture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MSC transplantion (Experimental): One group of glaucomatous patients will receive 10(6) autologous bone marrow-derived mesenchymal stem cells transplantation into their worst eyes, through an unique intravitreal injections, under anesthesia.
  Interventions: Procedure: Intravitreal transplantation of mesenchymal stem cell; Biological: Culture and isolation of autologous bone-marrow mesenchymal stem cells

INTERVENTIONS:
Procedure: Intravitreal transplantation of mesenchymal stem cell
Biological: Culture and isolation of autologous bone-marrow mesenchymal stem cells

SUMMARY:
Bone marrow-derived mesenchymal stem cells (MSC) therapy is a promising treatment for several degenerative diseases, including retinopathies and glaucoma, however no previous safety study involving humans has been conducted. The objective of this study is to evaluate effects of autologous bone marrow-derived MSC transplantation in the worst eye of 10 patients with legal bilateral blindness due to glaucoma. Primary outcome are types and severity of adverse effects. Secondary outcomes are changes in visual field, visual acuity, optical coherence tomography, and retinal ganglion cells function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Advanced Bilateral Open-Angle Glaucoma;
* Best corrected visual acuity less than 0,1 in the better eye;
* Social and cognitive ability to participate.

Exclusion Criteria:

* Severe systemic morbidities;
* Other ocular blind conditions associated;
* Impossibility in performing any of the proposed examinations.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayter S Paula, MD, Principal Investigator — Associate Professor
Locations (1):
- Ribeirão Preto Medical School, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Vilela CAP, Messias A, Calado RT, Siqueira RC, Silva MJL, Covas DT, Paula JS. Retinal function after intravitreal injection of autologous bone marrow-derived mesenchymal stromal cells in advanced glaucoma. Doc Ophthalmol. 2021 Aug;143(1):33-38. doi: 10.1007/s10633-021-09817-z. Epub 2021 Jan 19. PMID 33469852

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study requisits to enroll patients are too tight and some patients selected do not atend to all admision requisits like vision acuity worse than 20/100 in both eyes, absence of systemic comorbidities, etc.
Groups:
- MSC Transplantion: One group of glaucomatous patients will receive 10(6) autologous bone marrow-derived mesenchymal stem cells transplantation into their worst eye, through an unique intravitreal injections, under anesthesia.
  Intravitreal transplantation of mesenchymal stem cell
  Culture and isolation of autologous bone-marrow mesenchymal stem cells
Period: The First Patient Included at Study
Arm/Group | MSC Transplantion
Started | 1
Completed | 1
Not Completed | 0
Period: The Second Patient Included at Study
Arm/Group | MSC Transplantion
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- The First Patient Included at Study: On the thirtieth day after the vitreous injection a combined serous retinal detachment with proliferative vitreoretinopathy was noticed in patient 1 - promptly treated with a successful pars plana vitrectomy and silicone oil tamponade. At the final follow-up period (12 months), he remained with no retinal detachment and light perception vision.
Arm/Group | The First Patient Included at Study
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  Brazil | 2

OUTCOME MEASURES:

1. Primary Outcome: Type and Severity of Adverse Effects (AE) and Adverse Reactions (AR)
Description: Retinal detachment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | The First Patient Included at Study
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Changes in Visual Acuity
Time Frame: 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Visual Field
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Optical Coherence Tomography Parameters Related to Glaucoma
Time Frame: 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Retinal Ganglion Cells Function by ERG
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | The First Patient Included at Study
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The First Patient Included at Study (N=2)
Retinal detachment (Eye disorders) | 1 (1) — A combined serous retinal detachment with proliferative vitreoretinopathy was noticed in patient 1 - treated with vitrectomy and silicone oil tamponade. At the final follow-up period he remained with no retinal detachment and light perception vision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes